CLINICAL TRIAL: NCT06227130
Title: Does a 6-week Specially Designed Meditation, Mindfulness, and Yoga Program Reduce Perceived Stress in Resident General Practitioners? - A Randomized Controlled Trial With Crossover Design.
Brief Title: Meditation, Mindfulness, and Yoga to Reduce Perceived Stress in Resident Doctors - A Randomized Controlled Trial With Crossover Design
Acronym: MindYou
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Region Skane (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: Dnr 2023-05678-01
Record Dates: First submitted 2024-01-18; First posted 2024-01-26 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-04

CONDITIONS: Stress, Job
Keywords: yoga; mindfulness; meditation
MeSH Terms: conditions — Occupational Stress

STUDY DESIGN:
Intervention Model Description: Intervention group (IG) and waiting group (WG). IG will start with intervention program. After 6 weeks WG does the intervention program. PSS-questionnaire will be performed at baseline and after 6 weeks for both groups, and after 12 weeks for WG.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Experimental: Intervention A specially designed 6-week program incorporating meditation, mindfulness, and yoga, tailored to address specific challenges that resident doctors may face in their daily work. Each session lasts for about 20 minutes and the participant is encouraged to perform the session at least 3 times/week.
  Interventions: Behavioral: MindYou
- Waiting list (Active Comparator): The first 6 weeks of the study, the participants will be controls. During week 6-12 they will then perform the intervention according to the description above.
  Interventions: Behavioral: MindYou

INTERVENTIONS:
Behavioral: MindYou — A specially designed 6-week program incorporating meditation, mindfulness, and yoga, tailored to address specific challenges that resident doctors may face in their daily work.

SUMMARY:
General practitioners perceive their work as meaningful. However, according to a report from the Swedish Medical Association in 2022, about a quarter had considered leaving the profession altogether and nearly half had considered changing workplaces or reducing their working hours during the past 12 months. Several studies on mindfulness, yoga and meditation have shown effect on stress and burn out symptoms. The aim of the study is to investigate whether a specially designed 6-week program incorporating meditation, mindfulness, and yoga, tailored to address specific challenges that resident doctors may face in their daily work, can reduce perceived stress levels compared to a control group.

DETAILED DESCRIPTION:
The study is designed as a randomized controlled trial with a crossover design. The outcome measure is the level of stress assessed using the Perceived Stress Scale (PPS), Swedish version (PSS 14). Inclusion criteria are resident general practitioners in Skåne, within the preliminary catchment area of Malmö Trelleborg, who have experienced any form of stress symptoms they believe are related to their work. Participants will be recruited through an oral presentation during an educational seminar in spring 2024. Those who are interested will get a link to a webb-based questionnaire where they can fill in their informed consent and contact information. Participants will be randomised to intervention (I) or waiting list (C). The interventions lasts for 6 weeks and consists of a 6 different mindfulness/ meditation/yoga-sessions (lasting for 20 minutes each). The sessions will be sent to the participant on USB-stick or via webb-link. Each of the 6 sessions are tailored to address a specific challenge that resident doctors may face in their daily work. The preliminary themes that will be addressed are 'Handling Mistakes,' 'Letting Go of Work,' 'Setting Boundaries,' 'Taking Breaks,' 'Being Good Enough,' and 'Managing Work Stress. The participants are encouraged to perform the program at least 3 times/week. Both groups will fill in the PSS-questionnaire at study start and after 6 weeks.

The control group will start the intervention after the second questionnaire (week 7-12) and will fill out the PSS-questionnaire a third time after intervention completion. The results will be analysed according to intention to treat. The Mann-Whitney U-test will be used to compare whether there is a significant difference in the change of median values on PSS 14 between the intervention and control groups.

ELIGIBILITY:
Inclusion Criteria:

* Resident doctor in primary care having felt work related stress at any time

Exclusion Criteria:

* none

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2024-06-04 (Actual); Primary Completion 2025-02-14 (Actual); Study Completion 2025-04-01 (Actual)

PRIMARY OUTCOMES:
PSS14 | 12 weeks
  Self perceived stress According till PSS 14

CONTACTS AND LOCATIONS:
Overall Officials: Moa Wolff, Study Director — Lund University
Locations (2):
- Sweden (2):
  - Educational Meeting for Resident Physicians in Lund, Lund
  - Educational Meeting for Resident Physicians in Malmö, Malmo

IPD SHARING:
Plan to Share IPD: Undecided